CLINICAL TRIAL: NCT06575335
Title: Antibacterial Efficacy of Triphala Tooth Wipes in Reduction of Streptococcus Mutans Colonies in Differently Abled Children- A Randomized Clinical Trial
Brief Title: Triphala Tooth Wipes in Reduction of Streptococcus Mutans Colonies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sana Masood, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-3384/DUHS/Approval/2024/53
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Plaque Control
Keywords: differently abled; triphala; chlorhexidine; tooth wipes

STUDY DESIGN:
Intervention Model Description: The participants will be allocated in either of the two treatment arms through Sequentially Numbered, Opaque, Sealed Envelopes (SNOSE) by the principal investigator.
Who Masked: Participant, Outcomes Assessor
Masking Description: It will be a double-blinded study where the participants and the microbiologist will be unaware of the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triphala Tooth Wipe (Experimental): The three fruits of triphala (Terminalia chebula, Emblica officinalis and Terminalia bellerica) will be bought in powder form from an herbal drug vendor. A mixture will be made by combining equal proportion of all these three powders in distilled water. This will then be boiled till the volume reduces to 1/8th part of the initial volume. A sweetener will be added to the decoction followed by filtering using a white muslin cloth and then storing in a sterile amber-coloured glass bottle in a refrigerator. The decoction obtained will be subjected to dilution to obtain 0.6% concentration. This will then be used to impregnate the marketed tooth wipes fabric. The triphala tooth wipes will be cut, folded individually, and then packed. Each pack will contain 16 wipes.
  Interventions: Other: Triphala Tooth Wipe
- Chlorhexidine Tooth Wipe (Active Comparator): The commercially available mouthwash containing 0.2% chlorhexidine will be purchased from the market and will then be used to impregnate the marketed tooth wipes fabric. The chlorhexidine tooth wipes will be cut, folded individually, and then packed. Each pack will contain 16 wipes.
  Interventions: Other: Chlorhexidine Tooth Wipe

INTERVENTIONS:
Other: Triphala Tooth Wipe — The wipes will be used 1 hour after meal time, twice daily for consecutively 7 days. The sachet seal will be opened, the wipe will be taken out and rest of the sachet sealed again. The wipes will be unfolded and wrapped around index finger of right hand and all surfaces of child's teeth, gums, roof of the mouth and tongue will be cleaned.
  Arms: Triphala Tooth Wipe
Other: Chlorhexidine Tooth Wipe — Same as triphala tooth wipe
  Arms: Chlorhexidine Tooth Wipe

SUMMARY:
This double-blind randomized clinical trial will be conducted among differently abled institutionalized children. Sixty participants aged 6-12 years with mild intellectual disability (ID) will be enrolled in the study and divided into two treatment groups. The participants will be allocated in either of the two treatment arms through Sequentially Numbered, Opaque, Sealed Envelopes (SNOSE) by the principal investigator. One group will receive triphala tooth wipes and the other will be given chlorhexidine tooth wipes, both for 7 days twice a day. Supragingival plaque sample will be collected from the buccal surface of the permanent maxillary first molar and will be subjected to microbial analysis for Streptococcus mutans (S. mutans) colonies using colony-forming units per millilitre (CFU/ml).

The tooth wipes will be prepared by the principal investigator under supervision of Pharmacognosist at Department of Pharmaceutics and Pharmacognosy, University of Karachi, Pakistan.

DETAILED DESCRIPTION:
Preparation of Tooth Wipes:

Preparation of Triphala Tooth Wipes- The triphala decoction will be prepared by the principal investigator at Department of Pharmaceutics and Pharmacognosy, University of Karachi, Pakistan under the supervision of Pharmacognocist. The three fruits of triphala will be bought in powder form from an ayurvedic drug vendor. A mixture will be made by combining equal proportion of all these three powders in distilled water. This will then be boiled till the volume reduces to 1/8th part of the initial volume.

A sweetener will be added to the decoction followed by filtering using a white muslin cloth and then storing in a sterile amber-coloured glass bottle in a refrigerator. This will preserve its organoleptic properties and its quality for fourteen days.

The decoction obtained will be subjected to dilution to obtain concentration. This will then be used to impregnate the marketed tooth wipes fabric. The triphala tooth wipes will be cut, folded individually, and then packed using the wet wipes machine in a plain white packing by local pharmaceutical company. Each pack will contain 16 wipes.

Preparation of Chlorhexidine Tooth Wipes- The commercially available chlorhexidine mouthwash containing will be purchased from the market and will then be used to impregnate the marketed tooth wipes fabric. The chlorhexidine tooth wipes will be cut, folded individually, and then packed using the wet wipes machine in a plain white packing by local pharmaceutical company. Each pack will contain 16 wipes.

Data Collection:

Consent- Before initiation of the study, informed consent will be taken from the parent and/or guardian.

Proforma- The questionnaire will consist of their demographic details and Intelligence Quotient (IQ) score. The Streptococcus mutans count will be assessed on day 1 and day 7 of the intervention.

IQ Score- Mild ID having IQ score of 50-55 to ~70 will be part of the study. This IQ score will be provided by the institute's clinical psychologist who examines and score the patient as per American Association of Mental Deficiency (AAMD) criteria.

Microbial Analysis of the Plaque Sample- Under aseptic measures, the buccal surface of the permanent maxillary first molar will be dried with cotton swab and the supragingival plaque sample will be collected on baseline and Day 7 of the intervention prior to mealtime using sterile Gracey curette 1/2 by the principal investigator. Each of the specimen will be transferred into different sterile Eppendorf tubes having in 0.5 ml phosphate-buffered saline (PBS) to prevent cell rupture or shrinkage due to osmosis. The samples will be transported in an Ice Box. This will be cultured on the mitis salivarius agar with bacitracin in Dow Research Institute of Biotechnology and Biomedical Sciences (DRIBBS) by the microbiologist. The plates will be incubated anaerobically at 37◦C for 48 h for growth of S. mutans colonies will then be assessed at the baseline and on Day 7 of the intervention. The S. mutans count will be classified as Class 0 (none), Class 1 (<102), Class 2 (103-104) and Class 3 (10≥5) CFU/ml showing negligible, low, moderate and high caries susceptibility respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with informed consent
2. Children with mild intellectual disability as per American Association of Mental Deficiency (AAMD)
3. Age ranging from 6 to 12 years
4. One treatment group will be thirty children receiving triphala tooth wipes
5. The other treatment group will be thirty children receiving chlorhexidine tooth wipes

Exclusion Criteria:

1. Children who had received antibiotics within 3 months
2. Participants requiring urgent dental care during the period of study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Streptococcus mutans (S. mutans) count | The S. mutans count will be assessed at baseline and at day 8 of the intervention.
  Colony Forming Unit per millilitre (CFU/ml) classified as Class 0 (none), Class 1 (<102), Class 2 (103-104) and Class 3 (10≥5) CFU/ml showing negligible, low, moderate and high caries susceptibility

SECONDARY OUTCOMES:
Plaque Index | These counts will be assessed at baseline and at day 8 of the intervention.
  Silness and Loe Plaque Index: The score will range from 0 to 3; 0 (excellent), 0.1-0.9 (good), 1.0-1.9 (fair), and 2.0-3.0 (poor) oral hygiene.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Masood, BDS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dar-ul-Sukun, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
As it is confidential data, the investigators won't be sharing it.

REFERENCES:
- [Background] Mosaddad SA, Tahmasebi E, Yazdanian A, Rezvani MB, Seifalian A, Yazdanian M, Tebyanian H. Oral microbial biofilms: an update. Eur J Clin Microbiol Infect Dis. 2019 Nov;38(11):2005-2019. doi: 10.1007/s10096-019-03641-9. Epub 2019 Aug 1. PMID 31372904
- [Background] Lin Y, Chen J, Zhou X, Li Y. Inhibition of Streptococcus mutans biofilm formation by strategies targeting the metabolism of exopolysaccharides. Crit Rev Microbiol. 2021 Sep;47(5):667-677. doi: 10.1080/1040841X.2021.1915959. Epub 2021 May 3. PMID 33938347
- [Background] Baca P, Castillo AM, Liebana MJ, Castillo F, Martin-Platero A, Liebana J. Horizontal transmission of Streptococcus mutans in schoolchildren. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e495-500. doi: 10.4317/medoral.17592. PMID 22143733
- [Background] Lemos JA, Palmer SR, Zeng L, Wen ZT, Kajfasz JK, Freires IA, Abranches J, Brady LJ. The Biology of Streptococcus mutans. Microbiol Spectr. 2019 Jan;7(1):10.1128/microbiolspec.gpp3-0051-2018. doi: 10.1128/microbiolspec.GPP3-0051-2018. PMID 30657107
- [Background] Lin Y, Zhou X, Li Y. Strategies for Streptococcus mutans biofilm dispersal through extracellular polymeric substances disruption. Mol Oral Microbiol. 2022 Feb;37(1):1-8. doi: 10.1111/omi.12355. Epub 2021 Nov 22. PMID 34727414
- [Background] da Rosa SV, Moyses SJ, Theis LC, Soares RC, Moyses ST, Werneck RI, Rocha JS. Barriers in Access to Dental Services Hindering the Treatment of People with Disabilities: A Systematic Review. Int J Dent. 2020 Jul 23;2020:9074618. doi: 10.1155/2020/9074618. eCollection 2020. PMID 32774378
- [Background] Carniello V, Peterson BW, van der Mei HC, Busscher HJ. Role of adhesion forces in mechanosensitive channel gating in Staphylococcus aureus adhering to surfaces. NPJ Biofilms Microbiomes. 2020 Aug 21;6(1):31. doi: 10.1038/s41522-020-00141-z. PMID 32826897
- [Background] Deshpande MA, Baliga S, Thosar N, Rathi N, Jyothishi S, Deulkar PV, Bane SP. Evaluation of antibacterial efficacy of Triphala toothwipes on oral Streptococcus mutans count in intellectually disabled children. Spec Care Dentist. 2021 Sep;41(5):619-625. doi: 10.1111/scd.12597. Epub 2021 Apr 14. PMID 33852738
- [Background] Prakash S, Shelke AU. Role of Triphala in dentistry. J Indian Soc Periodontol. 2014 Mar;18(2):132-5. doi: 10.4103/0972-124X.131299. PMID 24872616
- [Background] Penmetsa GS, B V, Bhupathi AP, Rani P S, B V S, M V R. Comparative Evaluation of Triphala, Aloe vera, and Chlorhexidine Mouthwash on Gingivitis: A Randomized Controlled Clinical Trial. Contemp Clin Dent. 2019 Apr-Jun;10(2):333-337. doi: 10.4103/ccd.ccd_583_18. PMID 32308299
- [Background] Kaur S, Michael H, Arora S, Harkonen PL, Kumar S. The in vitro cytotoxic and apoptotic activity of Triphala--an Indian herbal drug. J Ethnopharmacol. 2005 Feb 10;97(1):15-20. doi: 10.1016/j.jep.2004.09.050. Epub 2004 Dec 25. PMID 15652269
- [Background] Biradar YS, Singh R, Sharma K, Dhalwal K, Bodhankar SL, Khandelwal KR. Evaluation of anti-diarrhoeal property and acute toxicity of Triphala Mashi, an Ayurvedic formulation. J Herb Pharmacother. 2007;7(3-4):203-12. doi: 10.1080/15228940802152869. PMID 18928142
- [Background] Phetkate P, Kummalue T, Rinthong PO, Kietinun S, Sriyakul K. Study of the safety of oral Triphala aqueous extract on healthy volunteers. J Integr Med. 2020 Jan;18(1):35-40. doi: 10.1016/j.joim.2019.10.002. Epub 2019 Oct 16. PMID 31680053
- [Background] Peterson CT, Denniston K, Chopra D. Therapeutic Uses of Triphala in Ayurvedic Medicine. J Altern Complement Med. 2017 Aug;23(8):607-614. doi: 10.1089/acm.2017.0083. Epub 2017 Jul 11. PMID 28696777
- [Background] Padiyar B, Marwah N, Gupta S, Padiyar N. Comparative Evaluation of Effects of Triphala, Garlic Extracts, and Chlorhexidine Mouthwashes on Salivary Streptococcus mutans Counts and Oral Hygiene Status. Int J Clin Pediatr Dent. 2018 Jul-Aug;11(4):299-306. doi: 10.5005/jp-journals-10005-1530. Epub 2018 Aug 1. PMID 30397374
- [Background] Selvi MM, Selvabalaji A, Chonat A, Ananthan V, Mani E, Chinnaswamy AD. A Comparative Evaluation of Antimicrobial Efficacy of Triphala and Calcium Hydroxide as Intracanal Medicament: An In Vitro Study. J Pharm Bioallied Sci. 2022 Jul;14(Suppl 1):S774-S780. doi: 10.4103/jpbs.jpbs_168_22. Epub 2022 Jul 13. PMID 36110780
- [Background] Ahmed S, Shahnawaz K, Mandal TK, Ghafir M, Gummaluri SS, Vishal G. Comparative Evaluation of Antimicrobial Efficacy of Herbal Formulations of Septilin and Triphala with Conventional 2% Chlorhexidine on Root Canal and Oral Commensal Bacteria using Kirby Bauer Method: An in-vitro Study. Contemp Clin Dent. 2022 Oct-Dec;13(4):383-388. doi: 10.4103/ccd.ccd_423_21. Epub 2022 Nov 8. PMID 36686996
- [Background] Kumari U, Zafar T, Shafqat S, Askary SH, Qasim M, Kamran MA, Baig EA, Shaikh AC, Qureshi A. Caries-affected dentin disinfection using Triphala, Indocyanine green, and Potassium Titanyl Phosphate laser and their effect on adhesive bond strength. Photodiagnosis Photodyn Ther. 2023 Mar;41:103257. doi: 10.1016/j.pdpdt.2022.103257. Epub 2022 Dec 30. PMID 36592785
- [Background] Waldron C, Nunn J, Mac Giolla Phadraig C, Comiskey C, Guerin S, van Harten MT, Donnelly-Swift E, Clarke MJ. Oral hygiene interventions for people with intellectual disabilities. Cochrane Database Syst Rev. 2019 May 31;5(5):CD012628. doi: 10.1002/14651858.CD012628.pub2. PMID 31149734
- [Background] McGrath C, Zhou N, Wong HM. A systematic review and meta-analysis of dental plaque control among children and adolescents with intellectual disabilities. J Appl Res Intellect Disabil. 2019 May;32(3):522-532. doi: 10.1111/jar.12561. Epub 2019 Feb 8. PMID 30734986
- [Background] Blot S. Antiseptic mouthwash, the nitrate-nitrite-nitric oxide pathway, and hospital mortality: a hypothesis generating review. Intensive Care Med. 2021 Jan;47(1):28-38. doi: 10.1007/s00134-020-06276-z. Epub 2020 Oct 16. PMID 33067640
- [Background] Biradar YS, Jagatap S, Khandelwal KR, Singhania SS. Exploring of Antimicrobial Activity of Triphala Mashi-an Ayurvedic Formulation. Evid Based Complement Alternat Med. 2008 Mar;5(1):107-13. doi: 10.1093/ecam/nem002. PMID 18317557
- [Background] Srinagesh J, Krishnappa P, Somanna SN. Antibacterial efficacy of triphala against oral streptococci: an in vivo study. Indian J Dent Res. 2012 Sep-Oct;23(5):696. doi: 10.4103/0970-9290.107423. PMID 23422630
- [Background] Shanbhag VK. Triphala in prevention of dental caries and as an antimicrobial in oral cavity- a review. Infect Disord Drug Targets. 2015;15(2):89-97. doi: 10.2174/1871526515666150513105009. PMID 25966965
- [Background] Pradeep AR, Suke DK, Martande SS, Singh SP, Nagpal K, Naik SB. Triphala, a New Herbal Mouthwash for the Treatment of Gingivitis: A Randomized Controlled Clinical Trial. J Periodontol. 2016 Nov;87(11):1352-1359. doi: 10.1902/jop.2016.130406. Epub 2016 Jul 21. PMID 27442086
- [Background] Mamgain P, Kandwal A, Mamgain RK. Comparative Evaluation of Triphala and Ela Decoction With 0.2% Chlorhexidine as Mouthwash in the Treatment of Plaque-Induced Gingivitis and Halitosis: A Randomized Controlled Clinical Trial. J Evid Based Complementary Altern Med. 2017 Jul;22(3):468-472. doi: 10.1177/2156587216679532. Epub 2016 Dec 8. PMID 27932522
- [Background] Bhattacharjee R, Nekkanti S, Kumar NG, Kapuria K, Acharya S, Pentapati KC. Efficacy of triphala mouth rinse (aqueous extracts) on dental plaque and gingivitis in children. J Investig Clin Dent. 2015 Aug;6(3):206-10. doi: 10.1111/jicd.12094. Epub 2014 May 22. PMID 24850703
- [Background] Naiktari RS, Gaonkar P, Gurav AN, Khiste SV. A randomized clinical trial to evaluate and compare the efficacy of triphala mouthwash with 0.2% chlorhexidine in hospitalized patients with periodontal diseases. J Periodontal Implant Sci. 2014 Jun;44(3):134-40. doi: 10.5051/jpis.2014.44.3.134. Epub 2014 Jun 5. PMID 24921057
- [Background] Tandon S, Gupta K, Rao S, Malagi KJ. Effect of Triphala mouthwash on the caries status. Int J Ayurveda Res. 2010 Apr;1(2):93-9. doi: 10.4103/0974-7788.64413. PMID 20814522
- [Background] Srinagesh J, Pushpanjali K. Assessment of antibacterial efficacy of triphala against mutans streptococci: a randomised control trial. Oral Health Prev Dent. 2011;9(4):387-93. PMID 22238738
- [Background] Saxena S, Lakshminarayan N, Gudli S, Kumar M. Anti Bacterial Efficacy of Terminalia Chebula, Terminalia Bellirica, Embilica Officinalis and Triphala on Salivary Streptococcus Mutans Count - A Linear Randomized Cross Over Trial. J Clin Diagn Res. 2017 Feb;11(2):ZC47-ZC51. doi: 10.7860/JCDR/2017/23558.9355. Epub 2017 Feb 1. PMID 28384980
- [Background] Bajaj N, Tandon S. The effect of Triphala and Chlorhexidine mouthwash on dental plaque, gingival inflammation, and microbial growth. Int J Ayurveda Res. 2011 Jan;2(1):29-36. doi: 10.4103/0974-7788.83188. PMID 21897640
- [Background] Baratakke SU, Raju R, Kadanakuppe S, Savanur NR, Gubbihal R, Kousalaya PS. Efficacy of triphala extract and chlorhexidine mouth rinse against plaque accumulation and gingival inflammation among female undergraduates: A randomized controlled trial. Indian J Dent Res. 2017 Jan-Feb;28(1):49-54. doi: 10.4103/0970-9290.203622. PMID 28393817
- [Background] Kayalvizhi G, Nivedha D, Sajeev R, Prathima GS, Suganya M, Ramesh V. Evaluating the Efficacy of Xylitol Wipes on Cariogenic Bacteria in 19- to 35-month-old Children: A Double-blind Randomized Controlled Trial. Int J Clin Pediatr Dent. 2018 Jan-Feb;11(1):13-17. doi: 10.5005/jp-journals-10005-1476. Epub 2017 Feb 1. PMID 29805228
- [Background] Goyal CR, Qaqish JG, Sharma NC, Warren PR, Cugini M, Thompson MC. Plaque removal efficacy of a novel tooth wipe. J Clin Dent. 2005;16(2):44-6. PMID 16170975
- [Background] Navya PN, Dhananjaya G, Chandra P. Efficacy of chlorhexidine wipes on colonization of Pseudomonas aeruginosa and Staphylococcus aureus in both ventilator and nonventilator patients in pediatric intensive care unit. J Indian Soc Pedod Prev Dent. 2020 Jul-Sep;38(3):289-292. doi: 10.4103/JISPPD.JISPPD_268_20. PMID 33004728
- [Background] Ikeda M, Miki T, Atsumi M, Inagaki A, Mizuguchi E, Meguro M, Kanamori D, Nakagawa K, Watanabe R, Mano K, Aihara A, Hane Y, Mutoh T, Matsuo K. Effective elimination of contaminants after oral care in elderly institutionalized individuals. Geriatr Nurs. 2014 Jul-Aug;35(4):295-9. doi: 10.1016/j.gerinurse.2014.03.003. Epub 2014 Apr 20. PMID 24755196
- [Background] Ryu M, Ueda T, Sakurai K. An Interprofessional Approach to Oral Hygiene for Elderly Inpatients and the Perception of Caregivers Towards Oral Health Care. Int Dent J. 2021 Aug;71(4):328-335. doi: 10.1016/j.identj.2020.12.003. Epub 2021 Feb 25. PMID 33642042
- [Background] Featherstone JDB, Crystal YO, Alston P, Chaffee BW, Domejean S, Rechmann P, Zhan L, Ramos-Gomez F. Evidence-Based Caries Management for All Ages-Practical Guidelines. Front Oral Health. 2021 Apr 27;2:657518. doi: 10.3389/froh.2021.657518. eCollection 2021. PMID 35048005
- [Background] Lee E, Park S, Um S, Kim S, Lee J, Jang J, Jeong HO, Shin J, Kang J, Lee S, Jeong T. Microbiome of Saliva and Plaque in Children According to Age and Dental Caries Experience. Diagnostics (Basel). 2021 Jul 23;11(8):1324. doi: 10.3390/diagnostics11081324. PMID 34441259
- [Background] Qudeimat MA, Alyahya A, Karched M, Behbehani J, Salako NO. Dental plaque microbiota profiles of children with caries-free and caries-active dentition. J Dent. 2021 Jan;104:103539. doi: 10.1016/j.jdent.2020.103539. Epub 2020 Nov 25. PMID 33248211
- [Background] Patil RU, Nachan VP, Patil SS, Mhaske RV. A clinical trial on topical effect of probiotics on oral Streptococcus mutans counts in children. J Indian Soc Pedod Prev Dent. 2021 Jul-Sep;39(3):279-283. doi: 10.4103/jisppd.jisppd_519_20. PMID 34810345
- [Background] Latifi-Xhemajli B, Rexhepi A, Veronneau J, Kutllovci T, Ahmeti D, Bajrami S. Streptococcus Mutans Infections in Infants and Related Maternal/Child Factors. Acta Stomatol Croat. 2021 Sep;55(3):308-315. doi: 10.15644/asc55/3/8. PMID 34658377